CLINICAL TRIAL: NCT03355027
Title: INvestigating the Lowest Threshold of Vascular bENefits From LDL Cholesterol Lowering With a PCSK9 mAb InhibiTor (Alirocumab) in Patients With Stable Cardiovascular Disease (INTENSITY-HIGH)
Brief Title: Investigating the Lowest Threshold of Vascular Benefits From LDL Cholesterol Lowering in Patients With Stable CV Disease
Acronym: INTENSITY-HIGH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: University of Cambridge (Other)
Responsible Party: Principal Investigator, Joseph Cheriyan, MD, Consultant Physician & Clinical Pharmacologist/Associate Lecturer, Cambridge University Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: INTENSITY-HIGH
Record Dates: First submitted 2017-10-06; First posted 2017-11-28 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Atherosclerosis; Cardiovascular Diseases
Keywords: Low Density Lipoprotein Cholesterol (LDL); PCSK9; Alirocumab; Flow Mediated Dilatation; Arterial Stiffness; Carotid Intima Media Thickness; Inflammation; Endothelial function; FDG PET-CT; PET-MR; Ezetimibe
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases; Inflammation | interventions — alirocumab; Ezetimibe; Tablets; Atorvastatin; Rosuvastatin Calcium; Simvastatin

STUDY DESIGN:
Intervention Model Description: Randomisation to be performed to a 1:1 ratio.
  Alirocumab treatment arm*:
  Alirocumab (150mg) & Statin (either: Simvastatin 80mg od, Rosuvastatin 20mg/40mg od or Atorvastatin 40/80mg od)
  *May be required to complete a 4 week washout period on a statin before entering the study: Simvastatin 80mg od, Rosuvastatin 20mg/40mg od or Atorvastatin 40/80mg od.
  Comparator treatment arm*:
  Ezetimibe (10mg) & Statin (either: Simvastatin 80mg od, Rosuvastatin 20mg/40mg od or Atorvastatin 40/80mg od)
  *May be required to complete a 4 week washout period on a statin before entering the study: Simvastatin 80mg od, Rosuvastatin 20mg/40mg od or Atorvastatin 40/80mg od.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Alirocumab Treatment Arm (Experimental): 30 patients with stable cardiovascular disease to receive Alirocumab 150mg & prescribed one of the following: Atorvastatin 40mg/80mg or Simvastatin 80mg or Rosuvastatin 20mg/40mg. Dosing and dispensing to be performed at V3, V4, V5 and V6.
  Interventions: Drug: Alirocumab 150 MG/ML; Drug: Atorvastatin 40Mg Tablet; Drug: Atorvastatin 80Mg Tablet; Drug: Rosuvastatin 20Mg Tablet; Drug: Rosuvastatin 40Mg Tablet; Drug: Simvastatin 80mg
- Comparator Treatment Arm (Active Comparator): 30 patients with stable cardiovascular disease to receive Ezetimibe 10mg & prescribed one of the following: Atorvastatin 40mg/80mg or Simvastatin 80mg or Rosuvastatin 20mg/40mg. Dosing and dispensing to be performed at V3, V4, V5 and V6.
  Interventions: Drug: Ezetimibe 10Mg Tablet; Drug: Atorvastatin 40Mg Tablet; Drug: Atorvastatin 80Mg Tablet; Drug: Rosuvastatin 20Mg Tablet; Drug: Rosuvastatin 40Mg Tablet; Drug: Simvastatin 80mg

INTERVENTIONS:
Drug: Alirocumab 150 MG/ML — Dosing to be performed by subcutaneous injection in clinic
  Other Names: Praluent
  Arms: Alirocumab Treatment Arm
Drug: Ezetimibe 10Mg Tablet — Patients will be instructed to take once daily at night.
  Other Names: Ezetrol
  Arms: Comparator Treatment Arm
Drug: Atorvastatin 40Mg Tablet — Patients will be instructed to take once daily at night. Atorvastatin will be the preferred statin option for those with eGFR < 60 ml/min/1.73m2. Patient may be required to complete a 4 week run-in period on a statin prior to entering the study (dependent on eligibility)
Drug: Atorvastatin 80Mg Tablet — Patients will be instructed to take once daily at night. Atorvastatin will be the preferred statin option for those with eGFR < 60 ml/min/1.73m2. Patient may be required to complete a 4 week run-in period on a statin prior to entering the study (dependent on eligibility)
Drug: Rosuvastatin 20Mg Tablet — Patients will be instructed to take once daily at night. Rosuvastatin only to be prescribed if atorvastatin and simvastatin are not previously tolerated. Patient may be required to complete a 4 week run-in period on a statin prior to entering the study (dependent on eligibility)
  Other Names: Crestor
Drug: Rosuvastatin 40Mg Tablet — Patients will be instructed to take once daily at night. Rosuvastatin only to be prescribed if atorvastatin and simvastatin are not previously tolerated. Patient may be required to complete a 4 week run-in period on a statin prior to entering the study (dependent on eligibility)
  Other Names: Crestor
Drug: Simvastatin 80mg — Patients will be instructed to take once daily at night. Patient may be required to complete a 4 week run-in period on a statin prior to entering the study (dependent on eligibility)

SUMMARY:
The INTENSITY-HIGH study aims to answer if there are any limits to LDL reduction in relation to benefiting vascular health, exploring the mechanisms by which secondary prevention in patients with established heart disease may benefit from even lower LDL levels. By using PCSK9 inhibitors such as Alirocumab, very low LDL cholesterol levels not previously encountered in statin trials, can be achieved in patients with established heart disease on top of intensive statin treatment.

This research is being carried out because it is unclear what the lowest threshold of LDL cholesterol should be to attain significant reductions in CV risk in stable cardiovascular patients. It is unknown whether there is a true limit of LDL cholesterol below which there is no further improvement in endothelial function in stable cardiovascular patients, and, whether this is associated with a reduction in markers of both systemic and vascular inflammation.

Defining this may help identify individuals from the general population who may benefit from more aggressive lipid lowering treatment than standard statin treatment in terms of CV morbidity and mortality.

This study will be conducted in patients with stable cardiovascular disease, where they will be randomized to receive either a combination of Alirocumab and statin, or Ezetimibe plus statin. 60 patients will be recruited to this single center, randomized, open label, parallel group, mechanistic physiological study which will be conducted at Cambridge University Hospitals NHS Foundation Trust. In order to be eligible for enrollment to the study, some patients may have to complete a 4 week washout period on a suitable statin therapy. The total study duration for each participant will be approximately 14 weeks, where a series of non-invasive vascular studies and medical imaging assessments which will be conducted to observe vascular/systemic inflammation and to assess endothelial vascular function.This study is funded by JP Moulton Charitable Foundation.

DETAILED DESCRIPTION:
The INTENSITY-HIGH study primarily seeks to explore the physiological mechanisms (mainly using endothelial function and vascular imaging of inflammation) by which secondary prevention in patients with established cardiovascular disease may benefit from even lower LDL levels using PCSK9 therapies. This will then set the basis for potential changes to guidelines about what a "healthy cholesterol" level should be and the targets these should be achieving, or indeed if there is a plateau beyond which there is no further benefit on surrogates of CV disease.

Endothelial function can be measured in the peripheral vasculature in a number of different ways, which include venous occlusion plethysmography with intra-arterial infusions of acetylcholine, ischemia flow-mediated endothelium-dependent dilatation (FMD) of the brachial artery, reactive hyperemia peripheral arterial tonometry (RH-PAT) and others. A venous plethysmography measure of forearm blood flow to intra-arterial acetylcholine infusion is the most sensitive and direct measurement of endothelium release of nitric oxides, but is more invasive than other techniques. FMD is non-invasive and measures changes in the brachial artery to ischemia. It is acknowledged that whilst FMD has a larger coefficient variation and is more technician dependent, it is more patient-friendly in that it is of shorter duration procedure wise, is non-invasive and is repeatable over a short period; therefore we have employed this technique in this study to improve chances of patient acceptability. RH-PAT is an alternative non-invasive assessment which measures volume changes at the fingertip (a surrogate of reactive hyperemia), is easy to implement and is not operator dependent. However, as yet it remains not well validated. Therefore, flow mediated dilatation has been selected for this study.

Metabolically active inflammatory cells utilize more glucose than non-activated cells, and the degree of metabolic activity can be measured using 18-fluorodeoxyglucose positron emission tomography/computed tomography (FDG-PET/CT). Cellular FDG uptake is largely irreversible and correlates with glucose usage and macrophage numbers in both tumor cells and atherosclerotic plaques [38, 39]. FDG PET imaging has been successfully used to determine culprit plaques responsible for TIA and stroke [4042]. The signal has also been shown to be responsive to therapy, with clear reductions in FDG uptake noted in both humans and animal models of atherosclerosis [43, 44]. In addition, very recently, it has been shown that FDG-PET/CT is a reliable technique to assess changes in plaque structure with good reproducibility [40]. Taken together, these findings suggest a role for FDG PET/CT imaging in the assessment of the antiinflammatory potential of novel compounds such as PCSK9 therapies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with high risk CVD with LDL-Cholesterol ≤ 4.0mmol* OR patients with very high risk CVD with LDL-Cholesterol ≤3.5mmol/l**
* Male or female patients over 40 years of age inclusive at screening, with a body weight ≥ 45kg and BMI ≥ 18 - ≤ 40kg/m2
* Palpable brachial arterial pulse, as per study team assessment
* History of stable CV disease, defined as previous myocardial infarction (STEMI or NSTEMI), angioplasty, documented CAD (Stress echo, CT coronary angiography or invasive angiography), stroke, TIA or peripheral vascular disease without a recent event in the last 6 months (i.e. acute coronary syndrome, unstable angina, CABG, PCI, stroke, MI, carotid endarterectomy)
* Stable 'suitable statin therapy' over the last 6 weeks as defined by a "statin equivalent" of Simvastatin 80mg od, Rosuvastatin 20mg/40mg od or Atorvastatin 40/80mg od. If not on stable statin therapy, a willingness to commence statin therapy or, if already on statin therapy, a willingness to increase statin therapy to fit the "statin equivalent" dose required in the study (as open label therapy) during run-in period
* Patients not taking Ezetimibe, or, if on Ezetimibe willingness to be washed out prior to randomisation

High risk is defined as a history of any of the following: acute coronary syndrome (such as myocardial infarction or unstable angina requiring hospitalisation), coronary or other arterial revascularisation procedures, chronic heart disease, ischaemic stroke, peripheral arterial disease.

Very high risk is defined as recurrent cardiovascular events or cardiovascular events in more than 1 vascular bed (that is, polyvascular disease).

Exclusion Criteria:

* Uncontrolled hypertension BP > 180/110 mmHg on repeated measurements
* Fasting hypertriglyceridemia with fasting TG>10 mmol/L at screening
* Pregnancy or combined oral contraceptive pill or hormone replacement therapy or childbearing potential
* Any concomitant condition that, at the discretion of the investigator, may affect the participant's ability to complete the study
* Any known sensitivity to Alirocumab or monoclonal antibodies
* Patients with history of hypersensitivity reactions to any of the study drugs
* History of significant LFT's (3xULN ALT or AST elevation) by previous statin treatment
* History of previous myositis associated with statin treatment (i.e. myalgias or asymptomatic CK elevation > 5 x ULN)
* Type 1 or Type 2 diabetes, which is insulin dependent or on oral hypoglycaemics/diet with HbA1c (DCCT) > 8% (OR HbA1c (IFCC) > 64mmol/mol) at screening. Please note: fasting glucose to be checked again at first FDG-PET/CT scan, and if glucose > 11mol/L at that visit, patients will be excluded from the study
* History of any acute CV event within 6 months prior to the screening period
* Rheumatoid arthritis, connective tissue disorders and other conditions known to be associated with active chronic inflammation (e.g. Inflammatory Bowel Disease)
* Untreated hypothyroidism, known autoimmune myositis
* Patients with CKD (defined as eGFR < 30 ml/min/1.73m2) at baseline will be excluded from the study
* Participant in a previous research study in the last 3 years which involved exposure to significant ionising radiation (i.e. cumulative research radiation dose > 5 mSv)
* History of malignancy within the past 5 years (with the exception of localised carcinoma of the skin that has been resected for cure)
* History of alcohol/drug abuse or dependence within 6 months of the study, screening visit 1
* Use of systemic corticosteroids at the time of scanning or a period of 2 weeks prior to screening visit
* Lack of ability to provide informed consent
* An unwillingness for female patients of childbearing potential to use an effective form of contraception (see section 12.2.3)
* Treatment with medications that result in significant drug to drug interactions with study medications. Assignment to a specific statin will be allowed prior to randomisation on a case-to-case basis dependent on the interactions with concomitant medications

Inclusion/Exclusion Criteria for INTENSITY-HIGH PET/MR sub-study (optional)

* Patient meets Inclusion/Exclusion criteria for INTENSITY HIGH
* Patient who fulfills the local imaging centre requirements for being scanned in the PET/MR machine will be enrolled
* Patient is willing to consent to participate in the sub-study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Vascular inflammation (Standard Uptake Value) - Carotid artery | 8 weeks
  Change in vascular inflammation in the carotid artery between Alirocumab and Ezetimibe treatment regimes (Vascular inflammation will be quantified by calculating the Standard Uptake Value [SUV])
Vascular inflammation (Tissue to Background Ratio TBR) - Carotid artery | 8 weeks
  Change in vascular inflammation in the carotid artery between Alirocumab and Ezetimibe treatment regimes (Vascular inflammation will be quantified by calculating the Tissue to Background Ratio [TBR])
Vascular inflammation (Standard Uptake Value) - Aortic artery | 8 weeks
  Change in vascular inflammation in the aortic artery between Alirocumab and Ezetimibe treatment regimes (Vascular inflammation will be quantified by calculating the Standard Uptake Value [SUV])
Vascular inflammation (Tissue to Background Ratio TBR) - Aortic artery | 8 weeks
  Change in vascular inflammation in the aortic artery between Alirocumab and Ezetimibe treatment regimes (Vascular inflammation will be quantified by calculating the Tissue to Background Ratio [TBR])

SECONDARY OUTCOMES:
Endothelial-dependent vasodilatation (as measured by Flow Mediated Dilatation using high-resolution vascular ultrasound) | 8 weeks
  Comparing the effects of Alirocumab or Ezetimibe treatment regimes on Flow Mediated Dilatation (a surrogate of endothelial-dependent vasodilatation)
Endothelial-independent vasodilatation (as measured by Flow Mediated Dilatation using high-resolution vascular ultrasound) | 8 weeks
  Comparing the effects of Alirocumab or Ezetimibe treatment regimes on sublingual glyceryl trinitrate (GTN) response to Flow Mediated Dilatation (a surrogate of endothelial-independent vasodilatation)
Augmentation index (an indicator of arterial stiffness) | 8 weeks
  Change in Augmentation Index between visits and between Alirocumab or Ezetimibe treatment regimes
Pulse wave velocity | 8 weeks
  Change in aortic Pulse Wave Velocity between visits and between Alirocumab or Ezetimibe treatment regimes
Carotid IMT | 8 weeks
  Change in Carotid IMT between visits and between Alirocumab or Ezetimibe treatment regimes
Systemic inflammation (as measured by lipid profile) | 8 weeks
  Change in systemic inflammation (as measured by lipid profile) between visits and between Alirocumab or Ezetimibe treatment regimes
Systemic inflammation (as measured by hsCRP) | 8 weeks
  Change in systemic inflammation (as measured by hsCRP) between visits and between Alirocumab or Ezetimibe treatment regimes
Systemic inflammation (as measured by MMP9) | 8 weeks
  Change in systemic inflammation (as measured by MMP9) between visits and between Alirocumab or Ezetimibe treatment regimes
Systemic inflammation (as measured by IL2) | 8 weeks
  Change in systemic inflammation (as measured by IL2) between visits and between Alirocumab or Ezetimibe treatment regimes
Systemic inflammation (as measured by IL6) | 8 weeks
  Change in systemic inflammation (as measured by IL6) between visits and between Alirocumab or Ezetimibe treatment regimes
Systemic inflammation (as measured by oxLDL lipid subfractions) | 8 weeks
  Change in systemic inflammation (as measured by oxLDL lipid subfractions) between visits and between Alirocumab or Ezetimibe treatment regimes

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Cheriyan, MBChB, FRCP, MA, Principal Investigator — Cambridge University Hospitals NHS Trust; Michalis Kostapanos, MD, PhD, FRSPH, Principal Investigator — Cambridge University Hospitals NHS Trust
Locations (1):
- Addenbrooke's Hospital, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Only the minimum required participant identifiable information (name and contact details) will be provided to the research team for the purpose of arranging study visits and completing the informed consent process. All delegated research personnel that is responsible to conduct the data/statistical analysis will only analyse data that is anonymised of any patient identifiable data.

REFERENCES:
- [Derived] Cacciottolo PJ, Kostapanos MS, Hernan Sancho E, Pavey H, Kaloyirou F, Vamvaka E, Helmy J, Hubsch A, McEniery CM, Wilkinson IB, Cheriyan J. Investigating the Lowest Threshold of Vascular Benefits from LDL Cholesterol Lowering with a PCSK9 mAb Inhibitor (Alirocumab) in Patients with Stable Cardiovascular Disease (INTENSITY-HIGH): protocol and study rationale for a randomised, open label, parallel group, mechanistic study. BMJ Open. 2021 Apr 13;11(4):e037457. doi: 10.1136/bmjopen-2020-037457. PMID 33849844